CLINICAL TRIAL: NCT02004184
Title: Maintenance Pemetrexed Therapy After Induction Chemotherapy Versus Pemetrexed at Progression in Advanced Non-Small-Cell Lung Cancer: A Randomized Phase III Study
Brief Title: Pemetrexed in Advanced Non-Small-Cell Lung Cancer: at Progression vs Maintenance Therapy After Induction Chemotherapy
Acronym: IDA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor enrollment due to the introduction of immunotherapy
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/645; 2013-001237-41 (EudraCT Number)
Record Dates: First submitted 2013-11-19; First posted 2013-12-09 (Estimated); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Carcinoma, Non-small-cell Lung
Keywords: Pemetrexed; drug therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- maintenance pemetrexed (Experimental): maintenance pemetrexed immediately after induction chemotherapy
  Interventions: Drug: maintenance pemetrexed
- pemetrexed at progression (Active Comparator): observation and pemetrexed therapy at disease progression
  Interventions: Drug: pemetrexed at progression

INTERVENTIONS:
Drug: maintenance pemetrexed — 500 mg/m2 Body Surface Area is administered intravenously every 3 weeks
  Other Names: Alimta
  Arms: maintenance pemetrexed
Drug: pemetrexed at progression — 500 mg/m2 Body Surface Area is administered intravenously every 3 weeks
  Other Names: Alimta
  Arms: pemetrexed at progression

SUMMARY:
Non-small-cell lung cancer (NSCLC) accounts for a majority (approximately 85%) of lung cancer cases. Patients with localized disease can be cured through surgery, but only 20 % are operable.For the majority of patients with advanced disease, palliative cytotoxic chemotherapy remains the recommended therapy. Chemotherapy prolongs survival and improves quality of life.

The recommended first-line therapy is 4-6 courses of a platinum in combination with a third generation compound (e.g. gemcitabine, vinorelbine, docetaxel, pemetrexed, paclitaxel). After first-line therapy, it has been recommended to observe the patients and offer second-line chemotherapy at disease progression.

Regimens for second-line therapy include docetaxel or pemetrexed monotherapy. Pemetrexed is less toxic and superior to gemcitabine in non-squamous NSCLC, whereas docetaxel is the recommended second-line therapy in squamous cell carcinoma.

The results of the studies of maintenance pemetrexed therapy are encouraging; the observed survival benefit is clinically relevant and relatively large considering the poor survival in patients with advanced NSCLC. Furthermore, pemetrexed appears to be well tolerated. There are, however, several limitations to the studies that have been conducted: Relatively few elderly patients and no PS 2 patients were enrolled - and not all patients on the control-arms received pemetrexed at progression.

The overall aim of this study is to investigate whether immediate maintenance pemetrexed therapy prolongs survival compared to observation and pemetrexed therapy at progression in patients with advanced NSCLC. Furthermore, it will be explored whether patients with 'performance status' 2 and elderly ≥ 70 years tolerate and benefit from maintenance therapy; and what characteristics and blood biomarkers are associated with sensitivity and tolerability of such therapy.

DETAILED DESCRIPTION:
In previous studies without maintenance therapy, median overall survival (OS) for performance status (PS) 0-1 patients has been approximately 9 months, corresponding to 6 months from randomization in this study. We consider an improvement in overall survival of two months to be the minimum difference that will lead to routine use of maintenance pemetrexed in Norway. To demonstrate an improvement in median overall survival from 6 to 8 months with an α =0.05 and β =0.20, 198 evaluable patients are required on each arm. We expect a drop-out rate of maximum 10 %, and therefore intend to randomize a total of 436 patients (PS 0-1) - of which we expect 150 to be 70 years or older.

Sample size is calculated on PS 0-1 patients only. In addition, PS 2 patients will be randomized until the required number of PS 0-1 patients have been accrued. We estimate that a total of 100 PS 2 patients will be enrolled - sufficient for hypothesis-generating analyses of the benefit of maintenance therapy in elderly and PS 2 patients.

Based on experience from our previous studies we estimate that approximately 30% of patients will not complete or progress during induction chemotherapy; or be ineligible due deterioration of PS. Consequently, we need to include approximately 765 patients.

ELIGIBILITY:
Inclusion Criteria:

* Measureable disease according to the RECIST 1.1
* Previous radiotherapy is acceptable provided there are measurable, previously not irradiated lesions present
* Histologically or cytologically confirmed non-squamous non-small cell lung cancer
* Stage IIIB ineligible for curative therapy or stage IV disease
* ECOG Performance 0-2
* Adequate organ function defined as:

  1. Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤ 3 x upper limit of normal (ULN), or AST and ALT ≤ 5 x ULN if liver function abnormalities are due to underlying malignancy.
  2. Total serum bilirubin ≤ 1.5 x ULN
  3. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  4. Platelets ≥ 100 x 109/L
  5. Creatinine clearance > 45 ml/min
* Able to discontinue NSAIDs and ASA if reduced renal function
* All fertile patients should use safe contraception
* Written informed consent

Exclusion Criteria:

* prior systemic therapy for advanced non-small-cell lung cancer (including EGFR-TKI). Previous chemotherapy (e.g. adjuvant after surgery or for other cancer) is allowed if ≥ 3 months since the last course was administered.
* activating EGFR-mutation or ALK-translocation detected
* serious concomitant systemic disorders (for example active infection, unstable cardiovascular disease) that in the opinion of the investigator would compromise the patient's ability to complete the study or interfere with the evaluation of the efficacy and safety of the study treatment
* conditions - medical, social, psychological - which could prevent adequate information and follow-up
* clinically active cancer other than NSCLC
* known hypersensitivity or contraindications for the study drugs (vinorelbine, carboplatin, pemetrexed, B12, folate)
* pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
overall survival | 2 years
  All patients will be followed until death of any reason - assessed up to 24 months after inclusion in the study.

SECONDARY OUTCOMES:
progression free survival | 2 years
  From date of inclusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
Toxicity | 2 years
  All patients will be followed for 2 years (or until 1 month after the end of study therapy if study therapy is discontinued before 2 years after study inclusion).
Health related quality of life | 2 years
  All patients will be followed until discontinuation of study therapy - up to 24 months after inclusion in the study.

OTHER OUTCOMES:
Overall survival in elderly and PS 2 patients | 2 years
  All patients will be followed until death of any reason - assessed up to 24 months after inclusion in the study.
Associations between clinical characteristics and blood biomarkers - and outcomes of therapy | 2 years
  All patients will be followed until death of any reason - assessed up to 24 months after inclusion in the study.
Toxicity in elderly and PS 2 patients | 2 years
  All patients will be followed for 2 years (or until 1 month after the end of study therapy if study therapy is discontinued before 2 years after study inclusion).
Health related quality of life in elderly and PS 2 patients | 2 years
  All patients will be followed until discontinuation of study therapy - up to 24 months after inclusion in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn H Grønberg, MD PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Halvorsen TO, Stokke K, Killingberg KT, Raj SX, Sorhaug S, Brustugun OT, Flotten O, Helbekkmo N, Hornslien K, Madebo T, Fluge S, Gronberg BH. Randomized phase III trial comparing switch-maintenance pemetrexed with observation followed by pemetrexed at progression in advanced NSCLC. Acta Oncol. 2020 Sep;59(9):1051-1057. doi: 10.1080/0284186X.2020.1778179. Epub 2020 Jun 16. PMID 32543258
- [Derived] Stokke K, Sandvei MS, Gronberg BH, Slaaen M, Killingberg KT, Halvorsen TO. Prognostic Value of Post First-Line Chemotherapy Glasgow Prognostic Score in Advanced Non-Small Cell Lung Cancer. Clin Med Insights Oncol. 2022 Mar 22;16:11795549221086578. doi: 10.1177/11795549221086578. eCollection 2022. PMID 35342321